CLINICAL TRIAL: NCT04118283
Title: Improving the Assessment and Treatment of Chronic Pain in Veterans With Serious Mental Illness
Brief Title: Assessment and Treatment for Chronic Pain in Veterans With Serious Mental Illness
Acronym: CPSMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Maryland Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3069-W; 1IK2RX003069-01A2 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Schizophrenia; Psychotic Disorders; Bipolar Disorder; Affective Disorders, Psychotic
Keywords: Veterans; chronic pain; psychotic disorders; affective disorders, psychotic; cognitive behavioral therapy; ecological momentary assessment
MeSH Terms: conditions — Chronic Pain; Schizophrenia; Psychotic Disorders; Bipolar Disorder; Affective Disorders, Psychotic | interventions — Cognitive Behavioral Therapy; Health

STUDY DESIGN:
Intervention Model Description: This study involves a pilot randomized controlled trial (RCT) with 45 Veterans with co-occurring SMI and chronic musculoskeletal pain to examine feasibility and acceptability of Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) and preliminarily evaluate participant responses to intervention. The first 45 Veterans who pass screening will be enrolled and randomized to study condition on a rolling basis. Participants will be randomly assigned at a 2:1 ratio to CBT-CP:Health & Wellness using permuted block randomization with randomly varying block sizes. Veterans will be randomly assigned to either CBT-CP (n = 30) or a manualized Health & Wellness active control intervention (n = 15). Using an intent-to-treat framework, data will be collected from every participant during the one-week Ecological Momentary Assessment period (prior to RCT baseline assessment) and at baseline, post-treatment, and 3-month follow-up regardless of attendance in their assigned condition.
Who Masked: Outcomes Assessor
Masking Description: Data will be collected by experienced Research Assistants (Ras) who will receive in-person training on each assessment measure. All RAs involved in the research study will conduct baseline assessments. One RA will remain blind to study condition in order to complete post-treatment and follow-up assessments. A back-up RA supplied by the VISN 5 MIRECC will be trained to conduct assessments in case the blind assessor is unblinded or in need of assistance. If the study condition becomes known, the blind assessor will stop the assessment and either the back-up RA or study PI will finish the assessment(s).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavioral Therapy for Chronic Pain (Experimental): Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) will be conducted in accordance with the Cognitive Behavioral Therapy for Chronic Pain: Therapist Manual and the VA Evidence-Based Practice (EBP) roll-out training. CBT-CP consists of a 12-session protocol, including an initial assessment session (BL assessment; Session 1), 10 content-specific sessions (pain education, goal-setting, cognitive and behavioral skill building; Sessions 2-11), and a booster session scheduled approximately one month after the final CBT-CP session (Session 12). Participants randomized to the CBT-CP condition (n = 30) will complete one 60-minute individual session per week. Each CBT-CP session will be led by a trained study interventionist using a manualized curriculum, following a basic structure including review of previous session material, introduction of new information or skills, and discussion of how to implement learned material into a home action plan.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Chronic Pain
- Health and Wellness (Active Comparator): Health & Wellness was developed by VISN 5 MIRECC investigators and consists of psychoeducation on topics related to physical and emotional wellbeing. Its structure is similar to CBT-CP (10 weekly individual 60-minute sessions, no booster session). Each Health & Wellness session will be led by a trained interventionist using a manualized curriculum that includes review of previous session material, introduction of new information, and discussion of a range of health-related topics (physical activity/exercise, nutrition/healthy eating, managing medications and side effects, and addictive behaviors (e.g., substance use, gambling, eating) that do not include pain. Typical sessions include discussion of the impact of the topic on overall health and well-being, identifying benefits and challenges to improving or maintaining health in that area, and strategies to address challenges in that area.
  Interventions: Behavioral: Health and Wellness

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Chronic Pain — Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) will be conducted in accordance with the Cognitive Behavioral Therapy for Chronic Pain: Therapist Manual and the VA Evidence-Based Practice (EBP) roll-out training. CBT-CP consists of a 12-session protocol, including an initial assessment session (BL assessment; Session 1), 10 content-specific sessions (pain education, goal-setting, cognitive and behavioral skill building; Sessions 2-11), and a booster session scheduled approximately one month after the final CBT-CP session (Session 12). Participants randomized to the CBT-CP condition (n = 30) will complete one 60-minute individual session per week. Each CBT-CP session will be led by a trained study interventionist using a manualized curriculum, following a basic structure including review of previous session material, introduction of new information or skills, and discussion of how to implement learned material into a home action plan.
  Other Names: CBT-CP
  Arms: Cognitive Behavioral Therapy for Chronic Pain
Behavioral: Health and Wellness — Health & Wellness was developed by VISN 5 MIRECC investigators and consists of psychoeducation on topics related to physical and emotional wellbeing. Its structure is similar to CBT-CP (10 weekly individual 60-minute sessions, no booster session). Each Health & Wellness session will be led by a trained interventionist using a manualized curriculum that includes review of previous session material, introduction of new information, and discussion of a range of health-related topics (physical activity/exercise, nutrition/healthy eating, managing medications and side effects, and addictive behaviors (e.g., substance use, gambling, eating) that do not include pain. Typical sessions include discussion of the impact of the topic on overall health and well-being, identifying benefits and challenges to improving or maintaining health in that area, and strategies to address challenges in that area.
  Other Names: H&W
  Arms: Health and Wellness

SUMMARY:
Chronic pain has a highly negative impact on Veterans, especially those with serious mental illness (SMI). Chronic pain leads to poorer mental health and physical functioning, and represents a critical obstacle to rehabilitation and recovery. Despite known high prevalence rates of chronic pain in SMI populations, there is little research to: a) evaluate nonpharmacological pain management strategies in this population, and b) examine directional relations between chronic pain and SMI symptoms. This study aims to address research and clinical gaps by: a) testing the feasibility and acceptability of Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) - a VA evidence-based psychotherapy for chronic pain - in Veterans with SMI, and b) better assessing the complex relation between chronic pain and psychiatric symptoms and their impact on functioning. Results from this study will inform us as to whether CBT-CP is feasible to implement, acceptable to Veterans with SMI, and worth examining in its standard or in an optimized form in a larger clinical trial.

DETAILED DESCRIPTION:
This research study will address critical gaps in our understanding and management of chronic musculoskeletal pain in Veterans with serious mental illness (SMI), addressing the following aims:

Aim 1: Complete a pilot randomized controlled trial (RCT) with 45 Veterans with co-occurring SMI and chronic musculoskeletal pain to examine feasibility and acceptability of CBT-CP and preliminarily evaluate participant responses to intervention.

Aim 1a (Primary): Determine feasibility by demonstrating adequate rates of recruitment and completion of and fidelity to the CBT-CP intervention as well as quality and acceptability of chosen assessments.

Aim 1b (Primary): Determine acceptability by obtaining favorable ratings from satisfaction questionnaires and interviews.

Aim 1c (Exploratory): Preliminarily evaluate participant responses to intervention by exploring changes in functioning and quality of life among Veterans randomized to the CBT-CP condition (n=30).

Aim 2: Determine the feasibility of collecting EMA data to examine the temporal relationships among mental health symptoms, pain severity, and health-related functioning. Data will be collected at baseline from the 45 Veterans in the Aim 1 RCT.

Aim 2b (Primary): Determine feasibility of this approach through adherence to the EMA call schedule and overall response rates.

Aim 2a (Exploratory): Explore relationships among mental health symptoms, pain severity, and health-related functioning captured in real time.

Aim 3: Complete a well-specified process evaluation to explore how to optimize CBT-CP for use in Veterans with SMI and chronic musculoskeletal pain in future clinical trials. This evaluation will integrate qualitative data from 15 interviews with Veterans in the CBT-CP condition, CBT-CP interventionist notes, and quantitative data from Aims 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Have a chronic musculoskeletal pain diagnosis
* Have a Defense and Veterans Pain Rating Scale (DVPRS) rating of 4 or greater for pain severity
* Meet criteria for an SMI diagnosis (schizophrenia, schizoaffective disorder, bipolar disorder) per medical record
* 18 years of age or older
* Enrolled in outpatient programming within the VA Maryland Health Care System at time of consent/study reenrollment
* Have regular access to a telephone
* Capacity to sign informed consent

Exclusion Criteria:

* Are engaging in moderate-to-severe substance use that would impact their ability to participate and/or would require a higher level of care (as determined by treating provider)
* Engagement in Cognitive Behavioral Therapy for Chronic Pain (CBT-CP), whether currently or in the past
* Have a current acute pain condition or limited mobility (i.e., unable to walk one city block) that would interfere with their ability to engage in CBT-CP interventions (e.g., activity pacing/walking program)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Participant Satisfaction Questionnaire (CSQ-8) | Participants will be assessed following completion of the study intervention, an expected average of 10 weeks
  The CSQ-8 contains eight Likert scale items that ask about quality of service received and if services have been helpful. Scores on the CSQ-8 range from 8 (lowest) to 32 (highest). This measure will be used to assess CBT-CP acceptability (Aim 1b).
Service Satisfaction Scale (SSS-30) | Participants will be assessed following completion of the study intervention, an expected average of 10 weeks
  The SSS-30 has 30 items that assess practitioner manner and skill, perceived outcome, office procedures, and accessibility. An overall score ranges from 30 (lowest) to 150 (highest). This measure will be used to assess CBT-CP acceptability (Aim 1b).
Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) Feasibility | Data will be gathered from each participant through intervention completion, an average of 10 weeks
  To examine feasibility, engagement and participation in CBT-CP will be tracked across four key objectives: 1) evaluation of recruitment and suitability of eligibility criteria (# consented divided by # approached; # randomized divided by # consented); 2) retention and adherence rates based on the percent who engaged in treatment (% of randomized who attend first 3 sessions) and mean number of sessions attended and treatment dropout percentages (# who dropped out prior to completing treatment divided by # who engaged); 3) outreach efforts (mean number of reminders and outreach contacts made for each participant); and 4) the mean (and SD) number of completed CBT-CP homework assignments, assessed weekly by CBT-CP interventionists.

SECONDARY OUTCOMES:
West Haven-Yale Multidimensional Pain Inventory (WHYMPI) - Interference | Participants will be assessed following completion of the study intervention, an expected average of 10 weeks
  The West Haven Yale Multidimensional Pain Inventory (WHYMPI) is a 52-item questionnaire providing a comprehensive assessment of components of the chronic pain experience that are helpful for the cognitive-behavioral conceptualization of chronic pain conditions. Each item is rated on a 7-point scale. The interference subscale will be used in this study and measures the impact of pain on functioning (household chores, outdoor work, recreation activities, social activities). An average score is calculated that ranges from 0 (no interference) to 6 (extreme interference). The WHYMPI has been used with a wide range of chronic pain populations and is sensitive to change following rehabilitative interventions. The WHYMPI is used as part of the CBT-CP assessment protocol.
Veterans RAND 36-item Health Survey (VR-36) | Participants will be assessed following completion of the study intervention, an expected average of 10 weeks
  The Veterans RAND 36-Item Health Survey (VR-36) is a 36-item questionnaire measuring health-related quality of life and 8 domains of health-related functioning (physical functioning, role limitations due to physical problems, role limitations due to emotional problems, bodily pain, general health perceptions, vitality, social functioning, and mental health). Items are scored on a 3- to 6-point scale and are summed to create each of the domain scores, ranging from 0 (worst health status) to 100 (best health status). The VR-36 demonstrated improved reliability, precision, and validity compared to the SF-36 and among persons with SMI.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Participants will be assessed following completion of the study intervention, an expected average of 10 weeks
  The WHODAS 2.0 is a 36-item questionnaire assessing health and disability across physical diseases and mental health disorders in both clinical and non-clinical settings and populations. Items are scored on a 5-point scale ranging from 0 (no difficulty) to 4 (extreme difficulty/cannot do) and are summed to create total (ranging from 0 to 144) and domain scores: understanding and communicating (ranging from 0 to 28); Getting around (ranging from 0 to 20); self-care (ranging from 0 to 16); getting along with people (ranging from 0 to 20); life activities (ranging from 0 to 32); and participating in society (ranging from 0 to 32). Higher scores for each domain indicate greater disability. Psychometric properties are excellent, with high internal consistency, test-retest reliability, a stable factor structure, good concurrent validity, and good sensitivity to change.
World Health Organization Quality of Life Scale (WHOQOL-BREF) | Participants will be assessed following completion of the study intervention, an expected average of 10 weeks
  The World Health Organization Quality of Life Scale (WHOQOL-BREF) is a 26-item questionnaire assessing four domains of quality of life: physical health, psychological well-being, quality of social relationships, and environmental quality. Items use different anchors but are rated on a scale from 1 to 5. Mean scores are calculated for each domain and then transformed to range from 0 (poorest quality of life) to 100 (best quality of life). Psychometric properties of the WHOQOL-BREF are excellent, with demonstrated high internal consistency, discriminant validity, and construct validity for general, mental health, and physical health populations. The WHOQOL-BREF is used as part of the CBT-CP assessment protocol.
West Haven-Yale Multidimensional Pain Inventory (WHYMPI) - Interference | Participants will be assessed a second time following completion of the study intervention, an expected average of 22 weeks.
  The West Haven Yale Multidimensional Pain Inventory (WHYMPI) is a 52-item questionnaire providing a comprehensive assessment of components of the chronic pain experience that are helpful for the cognitive-behavioral conceptualization of chronic pain conditions. Each item is rated on a 7-point scale. The interference subscale will be used in this study and measures the impact of pain on functioning (household chores, outdoor work, recreation activities, social activities). An average score is calculated that ranges from 0 (no interference) to 6 (extreme interference). The WHYMPI has been used with a wide range of chronic pain populations and is sensitive to change following rehabilitative interventions. The WHYMPI is used as part of the CBT-CP assessment protocol.
Veterans RAND 36-item Health Survey (VR-36) | Participants will be assessed a second time following completion of the study intervention, an expected average of 22 weeks.
  The Veterans RAND 36-Item Health Survey (VR-36) is a 36-item questionnaire measuring health-related quality of life and 8 domains of health-related functioning (physical functioning, role limitations due to physical problems, role limitations due to emotional problems, bodily pain, general health perceptions, vitality, social functioning, and mental health). Items are scored on a 3- to 6-point scale and are summed to create each of the domain scores, ranging from 0 (worst health status) to 100 (best health status). The VR-36 demonstrated improved reliability, precision, and validity compared to the SF-36 and among persons with SMI.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Participants will be assessed a second time following completion of the study intervention, an expected average of 22 weeks.
  The WHODAS 2.0 is a 36-item questionnaire assessing health and disability across physical diseases and mental health disorders in both clinical and non-clinical settings and populations. Items are scored on a 5-point scale ranging from 0 (no difficulty) to 4 (extreme difficulty/cannot do) and are summed to create total (ranging from 0 to 144) and domain scores: understanding and communicating (ranging from 0 to 28); Getting around (ranging from 0 to 20); self-care (ranging from 0 to 16); getting along with people (ranging from 0 to 20); life activities (ranging from 0 to 32); and participating in society (ranging from 0 to 32). Higher scores for each domain indicate greater disability. Psychometric properties are excellent, with high internal consistency, test-retest reliability, a stable factor structure, good concurrent validity, and good sensitivity to change.
World Health Organization Quality of Life Scale (WHOQOL-BREF) | Participants will be assessed a second time following completion of the study intervention, an expected average of 22 weeks.
  The World Health Organization Quality of Life Scale (WHOQOL-BREF) is a 26-item questionnaire assessing four domains of quality of life: physical health, psychological well-being, quality of social relationships, and environmental quality. Items use different anchors but are rated on a scale from 1 to 5. Mean scores are calculated for each domain and then transformed to range from 0 (poorest quality of life) to 100 (best quality of life). Psychometric properties of the WHOQOL-BREF are excellent, with demonstrated high internal consistency, discriminant validity, and construct validity for general, mental health, and physical health populations. The WHOQOL-BREF is used as part of the CBT-CP assessment protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Letitia Travaglini, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT04118283/ICF_000.pdf